CLINICAL TRIAL: NCT06543264
Title: Efficacy of Cryotherapy in Managing Chemotherapy-Induced Peripheral Neuropathy in Children With Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, Lecturer of Physical Therapy for Pediatrics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cryotherapy and Leukemia
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Single (Outcomes Assessor) Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (control group) and Group B (study group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Experimental): Cryotherapy (apparatus)
  Interventions: Device: Cryotherapy
- the control group (No Intervention): not received cryotherapy

INTERVENTIONS:
Device: Cryotherapy — Cryotherapy is a pain treatment that uses a method of localized freezing temperatures to deaden an irritated nerve. Cryotherapy is also used as a method of treating localized areas of some cancers (called cryosurgery), such as prostate cancer and to treat abnormal skin cells by dermatologists
  Arms: the study group

SUMMARY:
This study aimed to assess the efficacy of cryotherapy in controlling Peripheral Neuropathy in cancer children

DETAILED DESCRIPTION:
Peripheral neuropathy is a serious condition characterized by symmetrical, distal damage to the peripheral nerves that may be caused by several classes of drugs, including chemotherapeutic agents. Chemotherapy-induced peripheral neuropathy (CIPN) is an adverse effect estimated to occur in up to 40% of patients undergoing chemotherapy, with its incidence increasing in patients being treated with multiple agents. Pharmacists play a pivotal role in the prevention and management of CIPN by recommending evidence-based pharmacologic and non pharmacologic strategies appropriate for the individual patient.Peripheral neuropathy (PN) is a systemic disease characterized by symmetrical, distal damage to the peripheral nerves that negatively impacts patient quality of life (QOL). Prolonged symptoms associated with PN can cause pain, interfere with functional ability (e.g., dressing, driving, house-work), and disrupt emotional health.

ELIGIBILITY:
Inclusion Criteria:

1. Their age will ranging from eight to seventeen years.
2. Children participated in this study will from both sexes.
3. Children receiving chemotherapy as medical treatment protocol
4. All children have polyneuropathy caused by chemotherapy.

Exclusion Criteria:

1. Children with Epilepsy.
2. Children with blood clotting disorder.
3. Children have Open wounds / broken skin
4. Children with severe cardiac disease
5. Uncooperative patients.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction studies (NCS) | nerve conduction velocity for sensory ulnar nerve at day 0
  nerve conduction velocity for sensory ulnar nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory ulnar nerve at day 90
  nerve conduction velocity for sensory ulnar nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory sensory median nerve at day 0
  nerve conduction velocity for sensory median nerve
Nerve conduction studies (NCS) | nerve conduction velocity for sensory sensory median nerve at day 90
  nerve conduction velocity for sensory median nerve

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, PHD, Principal Investigator — South Valley University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No